CLINICAL TRIAL: NCT03201042
Title: Lyme Test Indication Combinations (LyTIC) Study
Acronym: LyTIC
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: Oxford Immunotec (Industry)
Responsible Party: Sponsor
Other Study IDs: L3
Record Dates: First submitted 2017-06-21; First posted 2017-06-28 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-06

CONDITIONS: Lyme Disease
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- 1a:Lyme patients- Erythema Migrans(EM)rash present: Patients with newly diagnosed Lyme disease based on the presence of a physician-documented EM rash. PCR, serology and Tcell based assay.
  Interventions: Diagnostic Test: PCR based assay; Diagnostic Test: Serology based assay; Diagnostic Test: Tcell based assay
- 1b:Lyme patients no typical EM: Patients documented symptoms of early Lyme disease, without a typical EM rash present, and the physician's intention to treat for Lyme disease. PCR, serology and Tcell based assay
  Interventions: Diagnostic Test: PCR based assay; Diagnostic Test: Serology based assay; Diagnostic Test: Tcell based assay
- Cohort 2: healthy controls: Patients drawn from Lyme disease non-endemic areas and subjects with known exposure to Lyme disease will be excluded. PCR, serology and Tcell based assay.
  Interventions: Diagnostic Test: PCR based assay; Diagnostic Test: Serology based assay; Diagnostic Test: Tcell based assay

INTERVENTIONS:
Diagnostic Test: PCR based assay — Whole blood specimens will be tested for the presence of Borrelia DNA by PCR in a two-step test (Imugen). In Cohort 1a and 1b. The first step tests for the presence of any Borrelia DNA. The second step is employed on positive samples and tests for the presence of either B. burgdorferi DNA or B. miyamotoi DNA. Positivity by PCR has a short but early window in the infection cycle for Borrelia burgdorferi and results may enable this window period and diagnosis rates to be better defined.
  In addition co-infection PCR analysis will be performed for the presence of Babesia, Anaplasma or Ehrlichia DNA (Imugen).
Diagnostic Test: Serology based assay — 1. The Imugen Lyme Antibody Analysis which includes immunoglobulin M (IgM),immunoglobulin G (IgG), and immunoglobulin A (IgA) antibody capture immunoassay and IgG and IgM based Western blots. In Cohort 1a and 1b.
  2. The Immunetics C6 Lyme ELISA assay.
  3. A 2-tier Lyme test performed and interpreted according to Centers for Disease Control (CDC) Guidelines
  4. A Rickettsia antibody test will be used to identify Spotted Fever and Typhus fever groups infections.
  Lyme test methodologies generally indicate a need to run a combination of tests in order to overcome limitations in either sensitivity or specificity of the various individual tests. Performance of all these tests on the same set of samples should enable both individual and combinatorial performance values to be calculated and compared.
Diagnostic Test: Tcell based assay — A research based ELISpot assay will be performed on peripheral blood mononuclear cells (PBMC) extracted from whole blood samples to test for presence of T cells activated against Borrelia antigens. Unlike serology based methods, this signal may not persist over extended periods of time in the absence of Borrelia antigens. The diagnostic window may be different for a test measuring adaptive immune response (i.e. T cells) and thus such test may identify patients with undetectable antibody response and may aid sensitivity of diagnosis.

SUMMARY:
To establish performance of individual tests and combinations of tests (serological, molecular and cellular tests) in early Lyme infection diagnosis

DETAILED DESCRIPTION:
The present study aims to investigate the performance characteristics of both established and new assays for Borrelia burgdorferi infection and to assess the relative performance of appropriate combinations of these tests. The study will also investigate the effect of the time course of the infection and its treatment on the outcomes for the various tests. Polymerase Chain Reaction(PCR), serology and T cell based tests will be performed. In addition, tests for Babesia, Anaplasma, Ehrlichia and Rickettsia will also be performed as these pathogens can be carried by the same tick that carries Borrelia and may result in coinfection.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1a (typical EM and intention to treat):

Inclusion

1. Documented new onset Lyme disease EM rash (single or multiple) with photographic evidence provided to Oxford Immunotec.
2. Patient must be able to provide blood sample at the initial visit (prior to treatment initiation) and subsequent samples according to the schedule.
3. Patients 5 years of age or older, with a minimum weight of 40 pounds.
4. Patient able to read English and to give consent to study participation.
5. If patient is younger than 18 years of age a legally authorized representative must provide consent.

Cohort 1b (no typical EM; Lyme disease symptoms; intention to treat):

Inclusion

1. Patients with suspected Lyme disease, based on physician's examination, where the physician has the intention to treat for Lyme disease (i.e. patients who following initial examination were prescribed treatment for Lyme disease).
2. Documented new onset of Lyme disease symptoms without a typical EM rash or with no rash. If a rash is present, photographic evidence must be provided.
3. Patient must be able to provide blood sample at the initial visit (prior to treatment initiation) and subsequent samples according to the schedule.
4. Patients 5 years of age or older, with a minimum weight of 40 pounds.
5. Patient able to read English and to give consent to study participation.
6. If patient is younger than 18 years of age a legally authorized representative must provide consent.

Cohort 2 (Healthy subjects):

Inclusion

1. Subjects 5 years of age or older, with a minimum weight of 40 pounds.
2. Subjects never diagnosed with any tick borne disease including Lyme disease
3. Subjects able to read English and to give consent to study participation.
4. If subject is younger than 18 years of age a legally authorized representative must provide consent.

Exclusion Criteria:

* Exclusion Cohort 1a (typical EM and intention to treat):

  1. Patients with Lyme-like symptoms lasting longer than 1 month prior to study enrolment.
  2. Patients receiving treatment for any tick borne disease (including Lyme disease) prior to enrolment.
  3. Patients who received a Lyme vaccination.
  4. Patients with anemia defined as a serum hemoglobin <10gm/dL.
  5. Patients who are participating in, or plan to participate in, any investigational drug study.
  6. Patients who are considered unsuitable for the study by the Investigator.

Cohort 1b (no typical EM; Lyme disease symptoms; intention to treat):

1. Patients with Lyme-like symptoms lasting longer than 1 month prior to study enrolment.
2. Patients receiving treatment for any tick borne disease (including Lyme disease) prior to enrolment.
3. Patients who received a Lyme vaccination.
4. Patients with anemia defined as a serum hemoglobin <10gm/dL.
5. Patients who are participating in, or plan to participate in, any investigational drug study.
6. Patients who are considered unsuitable for the study by the Investigator.

Cohort 2 (Healthy subjects):

Exclusion

1. Subjects with a history of tick bite
2. Subjects with past or current tick borne disease diagnosis
3. Subjects at risk for tick borne diseases including Lyme disease
4. Subjects residing in endemic regions for tick borne diseases: Connecticut, Delaware, Maine, Maryland, Massachusetts, Minnesota, New Hampshire, New Jersey, New York, Pennsylvania, Rhode Island, Vermont, Virginia and Wisconsin.
5. Subjects who have ever visited non-urban areas of endemic regions for tick borne diseases: Connecticut, Delaware, Maine, Maryland, Massachusetts, Minnesota, New Hampshire, New Jersey, New York, Pennsylvania, Rhode Island, Vermont, Virginia and Wisconsin.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 500 subjects aged 5 years or older.
Sampling Method: Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Sample Data Analysis | Tests at different time points post inital presentation will be evaluated through study completion, an average of 1 year.
  The results will be used to calculate performance, including sensitivity and specificity of the tests under evaluation. The utility of these tests at different time points post initial presentation will be evaluated.

CONTACTS AND LOCATIONS:
Locations (60):
- United States (60):
  - Paradigm Clinical Research, Redding, California
  - Coastal Connecticut Research, New London, Connecticut
  - Circle CARE Center, Norwalk, Connecticut
  - Orthopaedic Foundation for Active Lifestyles, Inc, Stamford, Connecticut
  - Delaware Integrated Medicine, Georgetown, Delaware
  - Eastern Research, Inc., Hialeah, Florida
  - South Florida Clinical Trials SFCT, A member of the Alliance, Inc., Hialeah, Florida
  - South Coast Research Center, Miami, Florida
  - Advance Clinical Research, Meridian, Idaho
  - Acadia Clinical Research, Bangor, Maine
  - Integrative Health Center of Maine, Portland, Maine
  - Centennial Medical Group, Eldridge, Maryland
  - Klein & Associates, MD, PA, Hagerstown, Maryland
  - MD Medical Research, Inc., Oxon Hill, Maryland
  - Rockville Internal Medicine Group, Rockville, Maryland
  - NECCR Primacare Research,LLC, Fall River, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Metromedic Walk In, New Bedford, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - NECCR Primacare Research, LLC, Westford, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Asthma and Allergy Institute of MI, Clinton Township, Michigan
  - Oakland Medical Research, Troy, Michigan
  - Pinnacle Research, Sartell, Minnesota
  - Andrea Gaito, Basking Ridge, New Jersey
  - MAffiliated Medical Associates, Florham Park, New Jersey
  - Modern Medical, Brooklyn, New York
  - Private Practice-Johnathan Liebowitz, Brooklyn, New York
  - NY Arthritis Clinic, Brooklyn, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Private Practice-David Wurwitz, Flushing, New York
  - Adirondack Medical Research Center, Glens Falls, New York
  - NYCT, A member of Alliance, Inc., New York, New York
  - Mid Hudson Medical Research, Newburgh, New York
  - John T. Mather Hospital, Port Jefferson, New York
  - Rapid Medical Research, Cleveland, Ohio
  - Buckeye Health and Research, Columbus, Ohio
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - Bally Medical Group, Barto, Pennsylvania
  - Boyertown Medical Assoc., Boyertown, Pennsylvania
  - Collegeville Family Practice, Collegeville, Pennsylvania
  - Brandywine Clinic, Downingtown, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Pediatric Medical Associates of NTN/ABG, East Norriton, Pennsylvania
  - Liberty Family Practice/Square 1, Erie, Pennsylvania
  - Detweiler Family Practice, Lansdale, Pennsylvania
  - Green and Seidner Family Practice, Lansdale, Pennsylvania
  - Suburban Research Assoc., Media, Pennsylvania
  - Brookside Family Practice and Pediatrics, Pottstown, Pennsylvania
  - Spring-Ford Family Practice, Royersford, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Ocean State Clinical Research, Lincoln, Rhode Island
  - NECCR Primacare Research, LLC, Portsmouth, Rhode Island
  - Atascosa Clinical Trial, Lytle, Texas
  - Brookside Family Health Care, Hinesburg, Vermont
  - Millennium Clincial Trials, Arlington, Virginia
  - Burke Internal Medicine, Burke, Virginia
  - The Education and Research Foundation, Inc., Lynchburg, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Exemplar Research, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No